CLINICAL TRIAL: NCT05252221
Title: Addiction Telemedicine Consultation in Primary Care: Increasing Access to Pharmacotherapy and Specialty Treatment for Alcohol Problems Via Telehealth
Brief Title: Alcohol Telemedicine Consultation in Primary Care (ATC)
Acronym: ATC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1564446; R01AA028211 (NIH)
Record Dates: First submitted 2022-01-28; First posted 2022-02-23 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder (AUD); Pharmacist-Patient Relations; Alcohol Problem
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual Care (UC) will consist of treatment as usual, standard and systematic alcohol screening as part of the "rooming" process conducted by medical assistants, and brief interventions and referrals to addiction treatment delivered by PCPs. PCPs can also prescribe the same AUD medications as those in the ATC arm.
- ATC Service (intervention) (Active Comparator): ATC components include in-exam-room, real-time videoconferencing or phone contact with the PCPs and their patients, asynchronous, rapid response consultation via email or phone. ATC consultants will offer a flexible service that includes:
  1. Direct patient contact, via video or telephone, during primary care visits
  2. Motivational Interviewing (MI) - informed facilitation of patient engagement in addiction treatment,
  3. Advice to PCP regarding patient-specific treatment options, including pharmacotherapy, addiction treatment, and combined treatments
  Interventions: Other: ATC Intervention

INTERVENTIONS:
Other: ATC Intervention — The ATC intervention offers convenient access to specialty consultation for PCPs and offers patients direct access to addiction treatment in a non-stigmatized primary care setting
  Arms: ATC Service (intervention)

SUMMARY:
This pragmatic, cluster-randomized trial in adult primary care clinics in a healthcare system with a diverse membership will examine the effectiveness of an innovative, multi-faceted intervention, the Addiction Telemedicine Consultant (ATC) service using clinical pharmacists to facilitate alcohol use problems and alcohol use disorder (AUD) pharmacotherapy and specialty addiction treatment entry.

DETAILED DESCRIPTION:
This study will examine the effectiveness of a multi-faceted intervention - the Addiction Telemedicine Consultant service, or "ATC," which consists of:

* A 1-hour information session for Primary Care Providers (PCP) about alcohol problems; including alcohol use disorder (AUD) and AUD pharmacotherapy, provided by the research team in collaboration with Kaiser Permanente Northern California (KPNC) addiction medicine and clinical pharmacy leadership. Along with a post session evaluation via survey monkey.
* PCP access to expert addiction medicine consultation by KPNC clinical pharmacists, via telephone, videoconference, and secure messaging - during primary care patient visits with the patient present, or asynchronously without the patient present.

  * Real-time, in-exam-room consultations may include clinical pharmacist assistance with patient assessment, psychoeducation, motivational interventions, and facilitation of patient engagement in addiction treatment.
  * Asynchronous consultations without the patient present may include clinical pharmacist advice regarding patient-specific treatment options, including pharmacotherapy, psychosocial treatment, and combined treatments,
* Ongoing technical assistance for PCPs, including coaching and troubleshooting on alcohol problems assessment and AUD medication prescribing and treatment entry facilitation, from the ATC consultants, as needed.

This study will use electronic health record (EHR) data to examine treatment arm effects on implementation outcomes and patient outcomes recorded during the course of regular clinical care, and health services utilization over two years. The study will accomplish this through the following specific aims:

Aim 1: To compare the ATC and Usual Care arms on implementation outcomes: AUD medication prescription order rates and specialty addiction treatment referrals over two years.

Aim 2: To compare the ATC and UC arms on patient outcomes: AUD medication fills, addiction treatment initiation, alcohol use (quantity/frequency), and services utilization over two years.

Aim 3: To understand characteristics associated with ATC implementation, and barriers and facilitators of AUD medication prescription. We will examine provider characteristics (including potential race/ethnic and gender disparities) associated with ATC implementation outcomes using EHR and semi-structured qualitative interviews with PCPs and explore how the different elements of ATC (video consult, telephone, and email) facilitate its implementation. Provider characteristics and EHR portions of this aim involve data only.

ELIGIBILITY:
Inclusion Criteria:

* Adult KPNC members who had a primary care visit in Oakland or San Francisco Medical Center between 01/01/2020 and 12/31/2021 (~250,000)
* PCPs working in Oakland and San Francisco Medical Centers (~300).
* Chief physicians, PCPs, and medical assistants working the intervention arm clinics (n~40 Key Informants).

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41843 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Implementation Outcomes | 2 years
  AUD Medication Prescription Rate
Implementation Outcomes | 2 years
  Rates of referrals to specialty addiction treatment
AUD Medication Fills | 2 years
  AUD Medication Fills
Addiction Treatment Initiation Rate | 2 years
  Addiction Treatment Initiation Rate
Alcohol use (quantity/frequency) | 2 years
  Alcohol use (quantity/frequency)
Rates of referral to specialty Addiction Medicine department | 2 years
  Specialty addiction treatment referrals
Rates of emergency department utilization in the intervention arms | 2 years
  Health Service Utilization
Rates of inpatient services utilization in the intervention arms | 2 years
  Health Service Utilization

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Sterling, DrPh, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente, Oakland, California
  - Kaiser Permanente, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metz VE, Leibowitz A, Satre DD, Parthasarathy S, Jackson-Morris M, Cocohoba J, Sterling SA. Effectiveness of a pharmacist-delivered primary care telemedicine intervention to increase access to pharmacotherapy and specialty treatment for alcohol use problems: Protocol for the alcohol telemedicine consult cluster-randomized pragmatic trial. Contemp Clin Trials. 2022 Dec;123:107004. doi: 10.1016/j.cct.2022.107004. Epub 2022 Nov 13. PMID 36379437